CLINICAL TRIAL: NCT01405755
Title: Partnering With Media and Vaccination Program to Improve Infant and Young Child Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Mexican National Institute of Public Health (Other Government)
Responsible Party: Principal Investigator, Edward Frongillo, Jr., Professor, University of South Carolina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00007388
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Infant and Young Child Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- National Vaccine Program Plus Radio (Experimental): Appropriate complementary feeding messages delivered using: (a) nurses during the 1st National Vaccination Week (NVW); and (b) radio.
  Interventions: Behavioral: Appropriate complementary feeding messages
- Comparison (no intervention) (No Intervention): No complementary feeding messages delivered.

INTERVENTIONS:
Behavioral: Appropriate complementary feeding messages — Messages delivered through National Vaccine Program and radio
  Arms: National Vaccine Program Plus Radio

SUMMARY:
Infant and young child feeding (IYCF) is a key determinant of under-nutrition and overweight in young children. In Mexico, breastfeeding extends well into the second half of infancy, but animal-source foods, cereals, and legumes are not regularly provided to the child by 9 mo. This study evaluates whether knowledge and practices about dietary diversity and food consistency can be improved using a two-component intervention strategy in semi-urban communities in Mexico. The two components will deliver appropriate complementary feeding messages using: (a) nurses during the 1st National Vaccination Week (NVW); and (b) radio messages and interviews. The intervention is evaluated using a cluster randomized design in small semi-urban communities in two states in Mexico with pre- and post-test questionnaires designed to assess changes in feeding behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with healthy children between 6 and 24 mo

Exclusion Criteria:

* None

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 420 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Provision of flesh-food or vitamin A-rich food | Change from baseline to 5 months
  Mothers provide at least one flesh-food (i.e., beef, chicken, fish, liver) or one vitamin A-rich fruit or vegetable in the previous day

SECONDARY OUTCOMES:
Provision of solid, semi-solid, or soft foods (i.e., not runny soups or broths) Provision of solid, semi-solid, or soft foods | Change from baseline to 5 months
  Mothers provide solid, semi-solid, or soft foods (i.e., not runny soups or broths) at least 1 meal/d (6-12 mo) or 2 meals/d (12-24 mo)

CONTACTS AND LOCATIONS:
Locations (1):
- Mexican National Institute of Public Health, Cuernavaca, Morelos, Mexico

REFERENCES:
- [Derived] Monterrosa EC, Frongillo EA, Gonzalez de Cossio T, Bonvecchio A, Villanueva MA, Thrasher JF, Rivera JA. Scripted messages delivered by nurses and radio changed beliefs, attitudes, intentions, and behaviors regarding infant and young child feeding in Mexico. J Nutr. 2013 Jun;143(6):915-22. doi: 10.3945/jn.112.169235. Epub 2013 Apr 24. PMID 23616510